CLINICAL TRIAL: NCT02477878
Title: A Phase I Study of Donor BPX-501 T Cell Infusion for Adults With Recurrent or Minimal Residual Disease Hematologic Malignancies Post-Allogeneic Transplant
Brief Title: Study of Gene Modified Donor T Cell Infusion in Patients With Recurrent Disease After Allogeneic Transplant
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-008
Expanded Access: NCT03639844 (No longer available)
Record Dates: First submitted 2015-05-18; First posted 2015-06-23 (Estimated); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Lymphoma; Multiple Myeloma; Hematologic Neoplasms
Keywords: Adult leukemias and myelodysplasia; Adult lymphomas; Adult multiple myeloma; allogeneic stem cell transplant; donor lymphocyte infusion
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Lymphoma; Multiple Myeloma; Hematologic Neoplasms; Anemia, Refractory, with Excess of Blasts | interventions — AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- BPX-501 and Rimiducid (Experimental): All subjects will receive 3 cycles of BPX-501 T cell infusions at escalating dose levels (DL). DL1 on Day 0, DL2 on Days 30 and 60. The first dose of BPX-501 T cells will occur ≥30 days after hematopoietic stem cell transplant (HSCT).
  Two doses of Rimiducid ( 0.1 mg/kg and 0.4 mg/kg) will be investigated for the treatment of aGvHD after BPX-501 T cell infusion.
  Interventions: Biological: BPX-501; Drug: Rimiducid

INTERVENTIONS:
Biological: BPX-501 — Biological: T cells transduced with CaspaCIDe suicide gene
Drug: Rimiducid — Rimiducid administered to treat GVHD
  Other Names: AP1903

SUMMARY:
A Phase I study of BPX-501 T cell infusion in adults with recurrent or minimal residual disease (MRD) hematologic malignancies post-allogeneic transplant. The treatment consists of increasing doses of BPX-501 T cell infusions to achieve a clinical response. Rimiducid will be investigated for the treatment of aGvHD after BPX-501 T cell infusion to determine a dose that can mitigate GvHD and preserve the graft versus leukemia effect.

DETAILED DESCRIPTION:
Unmanipulated donor lymphocyte infusion (DLI) is used after stem cell transplantation to treat and prevent relapse, to prevent infections and to establish full donor chimerism. The addition of mature T cells which exhibit a broad repertoire of T cell immunity against viral and cancer antigens, might provide a clinical benefit. However, an expected side effect of the presence of mature T cells is the potential occurrence of acute graft-versus-host disease (aGVHD). BPX-501 contains genetically modified donor T cells that have an inducible safety switch iCasp9 suicide gene. Evidence has emerged that escalating DLI has achieved higher clinical response rate with lower GVHD occurrence. Optimization of DLI dose and schedule as well as strategies of donor T-cell manipulation may lead to the consistent ability to separate GVHD from GvL (graft-versus-leukemia) activity and improve the safety of DLI treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged >18yrs and < 65yrs
2. Clinical diagnosis of one of the following adult hematological malignancies

   1. Leukemia
   2. Myelodysplastic Syndromes
   3. Lymphomas
   4. Multiple myeloma
   5. Other high-risk hematologic malignancies eligible for stem cell transplantation per institutional standard Life expectancy >10 weeks
3. Evidence of recurrent disease that presents > 100 days or minimal residual disease (MRD) that presents > 30 days after one of the following:

   1. Matched related HSCT
   2. Mismatched related HSCT
4. Signed patient informed consent;
5. A minimum genotypic identical match of 4/8 is required, as determined by high resolution typing, at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, and HLA- DRB1
6. Performance status: Karnofsky score > 50%
7. Subjects with adequate organ function as measured by:

   1. Bone marrow:

      * > 25% donor T-cell chimerism
      * ANC >1 x 10E9/L
   2. Cardiac: left ventricular ejection fraction at rest must be >45%.
   3. Hepatic: direct bilirubin ≤ 3 x upper limit of normal, or AST/ALT ≤ 5 x upper limit of normal
   4. Renal: creatinine ≤ 2x of ULN for age
   5. Pulmonary: FEV 1, FVC, DLCO (diffusion capacity) > 50% predicted (corrected for hemoglobin)

Exclusion Criteria:

1. ≥ Grade II acute GVHD or chronic extensive GVHD due to a previous allograft at time of screening;
2. Active CNS involvement by malignant cells;
3. Current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings). The principal investigator is the final arbiter of this criterion;
4. Positive HIV serology or viral RNA
5. Pregnancy (positive serum βHCG test) or breast-feeding;
6. Subjects of reproductive potential unwilling to use effective forms of birth control or abstinence for a year after transplantation;
7. Bovine product allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
BPX-501 Safety | Month 24
  To evaluate the safety of 2 stratified dose levels of BPX-501 T cell infusions based on patient-donor match in adult subjects with hematological malignancies
Rimiducid Safety | Month 24
  evaluate the safety of the infusion of escalating doses of dimerizer drug rimiducid (AP1903) in subjects who develop acute GvHD after BPX-501 infusion
GvHD | Month 24
  Assess incidence and severity of acute and chronic GvHD
Rimiducid Activity | Month 24
  Determine the effect of Rimiducid on mitigating GvHD
Rimiducid Efficacy | Month 24
  Assess time to resolution of GvHD after administration of Rimiducid

SECONDARY OUTCOMES:
Response Rate | Month 24
  Measure overall survival, disease free survival and response rates after BPX-501 infusion
Translational | Month 24
  Evaluate BPX-501 T cell function

CONTACTS AND LOCATIONS:
Overall Officials: Bellicum Pharmaceuticals, Study Director — Bellicum Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - BMT Program at Northside Hospital, Atlanta, Georgia
  - University of Kansas, Westwood, Kansas
  - Roswell Park, Buffalo, New York
  - Oregon Health & Science University, Portland, Oregon
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No